CLINICAL TRIAL: NCT07395583
Title: Efficacy of Eccentric Over Concentric Hamstring Exercises in Elite Male Footballers for Preventing Non-Contact Hamstring Injuries: A Randomized Controlled Trial
Brief Title: Preventing Non-Contact Hamstring Injuries in Elite Footballers: Eccentric vs Concentric Training
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emirates Health Services (EHS) (Other Government)
Collaborators: Lincoln University College Malaysia (Other)
Responsible Party: Principal Investigator, Gulab Kappattakath, Senior Physiotherapist, Emirates Health Services (EHS)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MOHAP/DXB-REC/S.O.O/No178/2025
Record Dates: First submitted 2026-01-26; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Long-Term Eccentric, Concentric & Combined Hamstring Training Improves Strength, May Cut Injury Risk, and Enhances Performance in Elite Male Football Players
Keywords: Eccentric hamstring training, Concentric hamstring training, combined eccentric and concentric hamstring training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ECCENTRIC HAMSTRING TRAINING (Experimental): Eccentric Training
  Barbell Romanian Deadlift:
  Stand hip-width apart with a slight knee bend. Hold the barbell shoulder-width apart, keep the spine neutral, and hinge at the hips to lower the barbell toward the shins. Engage the core, hamstrings, and glutes to return to standing. 3 sets × 10-12 reps.
  Nordic Hamstring Curl:
  Kneel with feet secured. Maintain a straight line from shoulders to knees and slowly lower the body under hamstring control. Use hands for support if needed and assist returning to start. 3 sets × 10-12 reps.
  Dumbbell Stiff-Leg Deadlift:
  Hold 10 kg dumbbells at the sides with minimal knee bend. Hinge at the hips, lowering the weights until a hamstring stretch is felt. Engage hamstrings and glutes to stand upright. 3 sets × 10-12 reps.
  Interventions: Other: Eccentric training + regular football practice
- CONCENTRIC HAMSTRING TRAINING (Experimental): Concentric Training
  Seated Leg Curl:
  Sit on the leg curl machine with feet shoulder-width apart and knees aligned with the machine hinge. Place the pad on the lower calf, engage the core, and keep the spine neutral. Pull the toes upward and curl the heels toward the glutes without arching the lower back. Slowly return to the starting position. 3 sets × 10-12 reps.
  Lying Leg Curl:
  Lie prone on the machine with feet hip-width apart and knees aligned with the hinge. Keep the core and glutes engaged, head neutral, and shoulder blades retracted. Curl the heels toward the glutes without lifting the hips or arching the back, then return slowly. 3 sets × 10-12 reps.
  Prone Hamstring Curl with Resistance Band:
  Lie prone with one end of a resistance band secured and the other around the ankle. Start with the knee extended and bend the knee against resistance, then return slowly. 3 sets × 10-12 reps.
  Along with regular football training.
  Interventions: Other: Concentric training + regular football practice
- COMBINED CONCENTRIC AND ECCENTRIC HAMSTRING TRAINING (Experimental): Barbell Romanian Deadlift: Stand hip-width with a slight knee bend, bar shoulder-width. Keep spine neutral, hinge at hips to lower the bar, then return using hamstrings and glutes. 3×10-12.
  Nordic Hamstring Curl: Kneel with feet secured, body straight. Slowly lower under control and assist back if needed. 3×10-12.
  Dumbbell Stiff-Leg Deadlift: Hold 10 kg dumbbells, minimal knee bend. Hinge at hips, lower until hamstrings stretch, then stand tall. 3×10-12.
  Seated Leg Curl: Sit with knees aligned, core engaged. Curl heels toward glutes and return slowly. 3×10-12.
  Lying Leg Curl: Lie prone with hips down and core tight. Curl heels toward glutes, then lower with control. 3×10-12.
  Prone Band Curl: Lie prone, band around ankle. Bend knee against resistance and return slowly. 3×10-12.
  Performed alongside regular football training.
  Interventions: Other: Eccentric training + regular football practice; Other: Concentric training + regular football practice
- CONTROL GROUP (No Intervention): Control (regular football training only)

INTERVENTIONS:
Other: Eccentric training + regular football practice — Eccentric Training
  Barbell Romanian Deadlift:
  Stand hip-width apart with a slight knee bend. Hold the barbell shoulder-width apart, keep the spine neutral, and hinge at the hips to lower the barbell toward the shins. Engage the core, hamstrings, and glutes to return to standing. 3 sets × 10-12 reps.
  Nordic Hamstring Curl:
  Kneel with feet secured. Maintain a straight line from shoulders to knees and slowly lower the body under hamstring control. Use hands for support if needed and assist returning to start. 3 sets × 10-12 reps.
  Dumbbell Stiff-Leg Deadlift:
  Hold 10 kg dumbbells at the sides with minimal knee bend. Hinge at the hips, lowering the weights until a hamstring stretch is felt. Engage hamstrings and glutes to stand upright. 3 sets × 10-12 reps.
  Along with regular football training.
  Arms: COMBINED CONCENTRIC AND ECCENTRIC HAMSTRING TRAINING; ECCENTRIC HAMSTRING TRAINING
Other: Concentric training + regular football practice — Concentric Training
  Seated Leg Curl:
  Sit on the leg curl machine with feet shoulder-width apart and knees aligned with the machine hinge. Place the pad on the lower calf, engage the core, and keep the spine neutral. Pull the toes upward and curl the heels toward the glutes without arching the lower back. Slowly return to the starting position. 3 sets × 10-12 reps.
  Lying Leg Curl:
  Lie prone on the machine with feet hip-width apart and knees aligned with the hinge. Keep the core and glutes engaged, head neutral, and shoulder blades retracted. Curl the heels toward the glutes without lifting the hips or arching the back, then return slowly. 3 sets × 10-12 reps.
  Prone Hamstring Curl with Resistance Band:
  Lie prone with one end of a resistance band secured and the other around the ankle. Start with the knee extended and bend the knee against resistance, then return slowly. 3 sets × 10-12 reps.
  Along with regular football training.
  Arms: COMBINED CONCENTRIC AND ECCENTRIC HAMSTRING TRAINING; CONCENTRIC HAMSTRING TRAINING

SUMMARY:
Football is a sport with a high risk of injury, and hamstring muscle injuries are among the most common problems faced by players. These injuries can reduce a player's performance, cause time away from training and matches, and place a burden on medical teams and clubs. Many training programs recommend eccentric hamstring exercises to prevent these injuries, but there is limited evidence comparing eccentric exercises with concentric exercises or a combination of both, especially in elite male football players.

The purpose of this study is to compare the long-term effects of three different hamstring strengthening programs-eccentric training, concentric training, and a combination of both-on preventing non-contact hamstring injuries in elite male footballers. Each training program will last for three months, and the players will be followed for a total period of 12 months. The study will look at how these programs affect hamstring injury prevention, muscle strength and performance, flexibility, recurrence of injuries, and players' psychological satisfaction.

The study is based on the following expectations:

A three-month eccentric hamstring strengthening program will lead to long-term improvements in reducing hamstring injuries, improving muscle performance and flexibility, lowering injury recurrence, and increasing psychological satisfaction over a 12-month period.

A three-month concentric hamstring strengthening program will also result in long-term improvements in injury prevention, muscle performance, flexibility, injury recurrence, and psychological satisfaction.

A combined program of eccentric and concentric hamstring strengthening over three months will produce significant long-term benefits in injury prevention, muscle performance, flexibility, injury recurrence, and psychological satisfaction.

There will be clear differences in outcomes between the eccentric, concentric, combined, and control groups over the 12-month follow-up period.

Participants will be divided into four groups (A, B, C, and D) based on the type of training they receive. The study will include young male professional football players aged 18 to 30 years from the UAE who are citizens or permanent residents. All participants must speak English, have at least one year of football playing experience, and must not have had any hamstring injury in the past six months. Players who are interested in participating and provide written informed consent will be included.

Players will be excluded if they have had a hamstring injury in the last six months, are female, are under 18 or over 30 years old, have restrictions in knee movement, have undergone previous hamstring surgery, are currently enrolled in another official rehabilitation program, or do not agree to participate in the study.

Group A participants will perform eccentric hamstring exercises, including Nordic hamstring curls, dumbbell stiff-leg deadlifts, and barbell Romanian deadlifts. Group B participants will perform concentric hamstring exercises such as seated leg curls, lying leg curls, and prone hamstring curls using resistance bands. Group C participants will perform a combination of both eccentric and concentric hamstring exercises. Group D participants will continue with their usual football training only and will not perform any additional hamstring-specific exercises.

Before each training session, all participants in Groups A, B, and C will complete a 10-minute warm-up, consisting of five minutes of cycling, three minutes of stretching, and two minutes of rope jumping. Each training session will last at least 30 minutes. The exercise groups will complete three additional training sessions per week alongside their regular football training for a total of 12 weeks.

The results of this study will help determine which type of hamstring training program is most effective in preventing non-contact hamstring injuries and improving physical and psychological outcomes in elite male football players.

DETAILED DESCRIPTION:
Background and Rationale Football is associated with one of the highest injury rates among competitive sports, with hamstring muscle injuries representing a major cause of time loss, reduced performance, and increased medical burden. Epidemiological evidence indicates that approximately 80% of hamstring injuries in football occur without direct contact, most commonly during high-speed running, sprinting, acceleration, deceleration, and sudden changes of direction. These injuries are associated with high recurrence rates and may significantly impact player availability and long-term athletic performance.

Hamstring muscle function plays a critical role in knee and hip stability, particularly during the terminal swing phase of sprinting when the hamstrings are subjected to high eccentric loads. Muscle weakness, fatigue, reduced flexibility, and imbalances between concentric and eccentric strength have been identified as key intrinsic risk factors for hamstring strain injuries in footballers.

Eccentric hamstring strengthening exercises-such as the Nordic hamstring exercise-are widely advocated for injury prevention due to their ability to increase muscle strength, fascicle length, and neuromuscular control. However, emerging evidence suggests that concentric strengthening and combined eccentric-concentric programs may also contribute to improved muscle performance and fatigue resistance. Despite extensive research on eccentric training, direct comparisons between eccentric, concentric, and combined hamstring strengthening programs in elite male football players remain limited, particularly with long-term follow-up across an entire competitive season.

Therefore, this randomized controlled trial aims to systematically evaluate and compare the long-term effectiveness of eccentric, concentric, and combined hamstring strengthening programs in preventing non-contact hamstring injuries, improving muscle performance and flexibility, reducing injury recurrence, and enhancing psychological satisfaction in elite male footballers.

Aim of the Study To compare the long-term effects of eccentric, concentric, and combined hamstring strengthening programs-each conducted over a three-month intervention period-on non-contact hamstring injury prevention, muscle performance, flexibility, injury recurrence, and psychological satisfaction in elite male football players over a 12-month follow-up period.

Specific Objectives

1. To evaluate changes in the incidence of non-contact hamstring injuries following eccentric, concentric, and combined hamstring strengthening programs.
2. To assess improvements in hamstring muscle performance and flexibility in response to different strengthening protocols.
3. To determine the recurrence rate of hamstring injuries during the 12-month follow-up period.
4. To assess psychological satisfaction and perceived sports performance among players undergoing each intervention.
5. To identify the most effective hamstring strengthening approach for injury prevention and performance enhancement in elite male footballers.

Hypotheses

1. A three-month eccentric hamstring strengthening program will produce significant long-term improvements in injury prevention, muscle performance, flexibility, reduced recurrence rates, and psychological satisfaction over a 12-month period.
2. A three-month concentric hamstring strengthening program will result in significant long-term improvements in the same outcome measures.
3. A combined eccentric and concentric hamstring strengthening program will yield significant long-term benefits across all outcome measures.
4. Significant differences will exist among eccentric, concentric, combined, and control groups with respect to injury incidence, muscle performance, flexibility, recurrence rates, and psychological satisfaction over the 12-month follow-up period.

Study Design This study is designed as a single-blind randomized controlled trial conducted over a 12-month period. Eligible participants will be randomly allocated into four intervention groups.

Study Setting The study will be conducted in collaboration with selected elite football clubs across the United Arab Emirates. All exercise interventions and injury management will be supervised by qualified physiotherapists at the Physiotherapy and Sports Medicine Center, Ras Al Khaimah.

Randomization and Blinding Randomization will be performed using an automated system by an independent individual not involved in the study. Participants will be allocated sequentially into one of four groups to ensure balanced distribution. Due to the nature of the interventions, the study will follow an open-label design; however, outcome assessors will remain blinded to group allocation to reduce assessment bias.

Intervention Groups Group A: Eccentric Training + Regular Football Training

Participants will perform:

* Nordic hamstring curls
* Dumbbell stiff-leg deadlifts
* Barbell Romanian deadlifts Group B: Concentric Training + Regular Football Training

Participants will perform:

* Seated leg curls
* Lying leg curls
* Prone hamstring curls with resistance bands Group C: Combined Eccentric and Concentric Training + Regular Football Training Participants will perform all exercises listed in Groups A and B. Group D: Control Group Participants will continue with regular football training only, without additional hamstring-specific exercises.

Training Protocol

* Frequency: 3 sessions per week
* Duration: Minimum of 30 minutes per session
* Intervention period: 12 weeks
* Warm-up (10 minutes):

  * 5 minutes cycling
  * 3 minutes stretching
  * 2 minutes rope jumping All sessions will be supervised to ensure safety and adherence. Outcome Measures Primary Outcome
* Incidence of non-contact hamstring injuries Secondary Outcomes
* Hamstring flexibility (Sit-and-Reach Test, Active Knee Extension Test)
* Muscle performance (30-meter sprint time, vertical jump height)
* Injury recurrence rates
* Psychological satisfaction (Subjective Sports Performance Satisfaction Questionnaire) Assessments will be conducted at baseline, post-intervention (3 months), and at 6, 9, and 12 months.

Safety and Risk Management All interventions will be supervised by trained professionals. Participants will be monitored for adverse events, including muscle soreness, strain, or joint discomfort. Pain levels will be recorded using the Visual Analogue Scale, and thigh circumference will be measured to detect swelling. Immediate medical care will be provided if required.

Ethical Considerations Participation is voluntary, and players may withdraw at any time without penalty. Written informed consent will be obtained prior to participation. Confidentiality will be maintained through anonymized data storage and restricted access. Ethical approval will be obtained from relevant institutional and national ethics committees prior to study commencement.

Expected Outcomes It is anticipated that eccentric hamstring strengthening will demonstrate superior effectiveness in reducing non-contact hamstring injuries, improving flexibility, enhancing sprint performance, and increasing psychological satisfaction compared to concentric or combined programs. The findings are expected to inform evidence-based injury prevention strategies in elite football.

Dissemination of Results

Results will be disseminated through:

* PhD thesis submission
* Publication in Scopus-indexed journals
* National and international conferences
* Reports shared with participating clubs and sports authorities Project Duration Total duration: 12 months, including baseline assessment, intervention phase, follow-up assessments, and data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Players without any recent hamstring injuries (within the last 6 months) from certain clubs will be asked to join the trial.
* The trial will include young male professional football players aged 18-30 from the UAE who are citizens or permanent residents, English speaking, with no hamstring injuries in the last six months.
* Participants must have at least one year of experience playing football and be interested in participating in the study.

Exclusion Criteria:

* Players who have had hamstring injuries within the last 6 months, women, individuals under 18 and over 30 years old will be disqualified.
* Individuals who have any restrictions in exercising the knee, have undergone prior surgery on their hamstring, or decline to give written informed consent for the study are not eligible.
* Furthermore, we will not include player who are currently enrolled in other official rehabilitation programs.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 275 (Estimated)
Dates: Start 2026-02-07 (Estimated); Primary Completion 2027-02-07 (Estimated); Study Completion 2027-04-23 (Estimated)

PRIMARY OUTCOMES:
Incidence of non-contact hamstring injuries | 12 Months
  The incidence of non-contact hamstring strain injuries will be systematically monitored using a prospective time-loss injury surveillance model, ensuring consistent and accurate tracking throughout the study period. All reported injuries will undergo comprehensive clinical assessment and verification, after which they will be categorized according to their mechanism, with specific identification of non-contact injuries. To facilitate objective and reliable comparison across the four intervention groups, injury incidence will be standardized and expressed per 1,000 player-hours of exposure, providing a uniform metric that accounts for variations in individual training and match participation.

SECONDARY OUTCOMES:
Hamstring flexibility: Active Knee Extension | 12 Months
  In the Active Knee Extension (AKE) test, participants lie in a supine position with the hip flexed to 90 degrees. From this position, they are instructed to actively extend the knee as far as possible while maintaining the hip angle. Hamstring flexibility is quantified by measuring the deficit from full knee extension, expressed in degrees using a goniometer. A smaller extension deficit indicates greater hamstring flexibility.
Athletic Performance Assessment: 30-meter sprint test | 12 Months
  Sprint performance will be assessed using a 30-meter sprint test. Participants will be instructed to start from a standing position and sprint maximally over the designated distance. The total time taken to complete the 30 meters will be recorded in seconds using a stopwatch. Each participant will be given adequate rest between trials to minimize the effects of fatigue, and the best time recorded will be used for analysis. This test provides an objective measure of acceleration and sprinting ability.
Recurrence Rates of Hamstring Injury | 12 Months
  Recurrent hamstring injury is defined as a subsequent injury occurring at the same site within two months of a player returning to full participation following the index injury, as per the criteria described by Fuller et al. (2006).
Subjective Sports Performance Satisfaction | 12 Months
  Measured using the subjective rating scale by Nahum O. et al. (2016). Participants rate six items from 0 ("not at all satisfied") to 10 ("fully satisfied"), with the final performance score calculated as the mean of all items.
Hamstring flexibility: Sit-and-Reach test | 12 Months
  The Sit-and-Reach test is used to evaluate overall posterior chain flexibility, including the hamstrings, lower back, and gastrocnemius muscles. Participants sit with their legs fully extended and feet placed against a standardized sit-and-reach box. They are asked to reach forward as far as possible with both hands while keeping the knees extended. The distance reached beyond (or short of) the toes is recorded in centimeters, with higher values indicating greater flexibility.
Athletic Performance Assessment: Vertical jump | 12 Months
  Vertical jump performance will be assessed to evaluate lower-body explosive power. Participants will first measure their standing reach height while keeping both feet flat on the ground. They will then perform a maximal vertical jump, reaching as high as possible. The difference between the standing reach height and the maximum jump height will be calculated and recorded in centimeters. Multiple trials may be performed, with the highest jump used for final analysis.

IPD SHARING:
Plan to Share IPD: No
All data collected during the study will be recorded on designated research forms and handled with strict confidentiality. Each participant will be assigned a unique identification code, and no personal identifiers will be used in data analysis or reporting. Access to identifiable information will be restricted to the principal investigator and co-investigator only, who will be responsible for secure data storage. In accordance with ethical guidelines, participant data will not be disclosed, shared, or released to any unauthorized individual or third party.

REFERENCES:
- [Background] Coudeyre E, Pereira B, Lechauve JB, Girold S, Richard R, Dobija L, Lanhers C. Eccentric Muscle Strengthening Using Maximal Contractions Is Deleterious in Knee Osteoarthritis: A Randomized Clinical Trial. J Clin Med. 2024 Jun 4;13(11):3318. doi: 10.3390/jcm13113318. PMID 38893028
- [Background] Sato S, Yoshida R, Murakoshi F, Sasaki Y, Yahata K, Kasahara K, Nunes JP, Nosaka K, Nakamura M. Comparison between concentric-only, eccentric-only, and concentric-eccentric resistance training of the elbow flexors for their effects on muscle strength and hypertrophy. Eur J Appl Physiol. 2022 Dec;122(12):2607-2614. doi: 10.1007/s00421-022-05035-w. Epub 2022 Sep 15. PMID 36107233
- [Background] Ruas CV, Latella C, Taylor JL, Haff GG, Nosaka K. Comparison between Eccentric-Only and Coupled Concentric-Eccentric Contractions for Neuromuscular Fatigue and Muscle Damage. Med Sci Sports Exerc. 2022 Oct 1;54(10):1635-1646. doi: 10.1249/MSS.0000000000002959. PMID 36106831
- [Background] Magdalena PG, Bartlomiej B, Robert T, Malgorzata S, Hsing-Kuo W, Sebastian K. Acute fatigue-induced alterations in hamstring muscle properties after repeated Nordic hamstring exercises. Sci Prog. 2024 Apr-Jun;107(2):368504241242934. doi: 10.1177/00368504241242934. PMID 38592327
- [Background] Evangelidis PE, Shan X, Otsuka S, Yang C, Yamagishi T, Kawakami Y. Fatigue-induced changes in hamstrings' active muscle stiffness: effect of contraction type and implications for strain injuries. Eur J Appl Physiol. 2023 Apr;123(4):833-846. doi: 10.1007/s00421-022-05104-0. Epub 2022 Dec 10. PMID 36494585
- [Background] Corcelle B, Da Silva F, Monjo F, Gioda J, Giacomo JP, Blain GM, Colson SS, Piponnier E. Immediate but not prolonged effects of submaximal eccentric vs concentric fatiguing protocols on the etiology of hamstrings' motor performance fatigue. Eur J Appl Physiol. 2024 Nov;124(11):3215-3226. doi: 10.1007/s00421-024-05466-7. Epub 2024 Jun 7. PMID 38847870
- [Background] Ekstrand J, Bengtsson H, Walden M, Davison M, Khan KM, Hagglund M. Hamstring injury rates have increased during recent seasons and now constitute 24% of all injuries in men's professional football: the UEFA Elite Club Injury Study from 2001/02 to 2021/22. Br J Sports Med. 2022 Dec 6;57(5):292-8. doi: 10.1136/bjsports-2021-105407. Online ahead of print. PMID 36588400
- [Background] Montalvo AM, Schneider DK, Webster KE, Yut L, Galloway MT, Heidt RS Jr, Kaeding CC, Kremcheck TE, Magnussen RA, Parikh SN, Stanfield DT, Wall EJ, Myer GD. Anterior Cruciate Ligament Injury Risk in Sport: A Systematic Review and Meta-Analysis of Injury Incidence by Sex and Sport Classification. J Athl Train. 2019 May;54(5):472-482. doi: 10.4085/1062-6050-407-16. Epub 2019 Apr 22. PMID 31009238
- [Background] Ekstrand J, Askling C, Magnusson H, Mithoefer K. Return to play after thigh muscle injury in elite football players: implementation and validation of the Munich muscle injury classification. Br J Sports Med. 2013 Aug;47(12):769-74. doi: 10.1136/bjsports-2012-092092. Epub 2013 May 5. PMID 23645834
- [Background] Vatovec R, Kozinc Z, Sarabon N. Exercise interventions to prevent hamstring injuries in athletes: A systematic review and meta-analysis. Eur J Sport Sci. 2020 Aug;20(7):992-1004. doi: 10.1080/17461391.2019.1689300. Epub 2019 Nov 13. PMID 31680644
- [Background] Jones S, Almousa S, Gibb A, Allamby N, Mullen R, Andersen TE, Williams M. Injury Incidence, Prevalence and Severity in High-Level Male Youth Football: A Systematic Review. Sports Med. 2019 Dec;49(12):1879-1899. doi: 10.1007/s40279-019-01169-8. PMID 31452129
- [Background] Owoeye OBA, VanderWey MJ, Pike I. Reducing Injuries in Soccer (Football): an Umbrella Review of Best Evidence Across the Epidemiological Framework for Prevention. Sports Med Open. 2020 Sep 21;6(1):46. doi: 10.1186/s40798-020-00274-7. PMID 32955626
- [Background] Della Villa F, Buckthorpe M, Grassi A, Nabiuzzi A, Tosarelli F, Zaffagnini S, Della Villa S. Systematic video analysis of ACL injuries in professional male football (soccer): injury mechanisms, situational patterns and biomechanics study on 134 consecutive cases. Br J Sports Med. 2020 Dec;54(23):1423-1432. doi: 10.1136/bjsports-2019-101247. Epub 2020 Jun 19. PMID 32561515
- [Background] Petersen J, Thorborg K, Nielsen MB, Budtz-Jorgensen E, Holmich P. Preventive effect of eccentric training on acute hamstring injuries in men's soccer: a cluster-randomized controlled trial. Am J Sports Med. 2011 Nov;39(11):2296-303. doi: 10.1177/0363546511419277. Epub 2011 Aug 8. PMID 21825112
- [Background] Huang YL, Jung J, Mulligan CMS, Oh J, Norcross MF. A Majority of Anterior Cruciate Ligament Injuries Can Be Prevented by Injury Prevention Programs: A Systematic Review of Randomized Controlled Trials and Cluster-Randomized Controlled Trials With Meta-analysis. Am J Sports Med. 2020 May;48(6):1505-1515. doi: 10.1177/0363546519870175. Epub 2019 Aug 30. PMID 31469584